CLINICAL TRIAL: NCT00333086
Title: A PHASE II STUDY OF LETROZOLE IN PATIENTS WITH ADVANCED OR RECURRENT ENDOMETRIAL CANCER
Brief Title: A Study of Letrozole in the Treatment of Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345ADE03
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent and Metastatic Endometrial Cancer
Keywords: Endometrial Cancer; Aromatase inhibitor; Letrozole
MeSH Terms: conditions — Recurrence; Endometrial Neoplasms | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
Currently available treatments for endometrial cancer are associated with limited efficacy and significant toxicity. This study will assess the safety and efficacy of letrozole, an aromatase inhibitor, on endometrial cancer.

ELIGIBILITY:
Inclusion criteria

* Postmenopausal women with recurrent or metastatic adeno- or adenosquamous carcinoma of the endometrium
* No adjuvant therapy
* Up to one prior hormonal (progestin) therapy for advanced/metastatic disease allowed
* No chemotherapy for recurrence (adjuvant permitted)
* Unidimensionally measurable disease
* Good Health status 0-2 (Eastern Cooperatitve Oncology Group)
* No prior tamoxifen or aromatase inhibitor therapy
* No other concurrent anti-cancer treatment
* No metastases in the central nervous system

Exclusion criteria:

Additional protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rates (complete response, partial response, no change, progressive disease) measured by tumor marker assessments and radiologic imaging at week 12 then every 12 weeks x 1 year followed by every 16 weeks

SECONDARY OUTCOMES:
Duration of clinical response, time to progression of the disease, correlation of tumor response with pretreatment ER/PR status, histological grade and aromatase levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Heidelberg, Germany